CLINICAL TRIAL: NCT07230171
Title: Comparing the Efficacy and Safety of Conventional Therapy With Conventional Therapy Combined Esketamine in the Treatment of Fibromyalgia: A Multicenter Clinical Study
Brief Title: The Efficacy and Safety of Short Term S-ketamine Infusion as an Adjunctive Therapy in Patients With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Ditan Hospital (Other); Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-217-03-06
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia; Pregabalin; Esketamine
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin; Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Pregabalin and venlafaxine concomitant therapy
  Interventions: Drug: Pregabalin and venlafaxine concomitant therapy
- Treatment group (Experimental): Esketamine plus pregabalin and venlafaxine concomitant therapy
  Interventions: Drug: Esketamine plus pregabalin and venlafaxine concomitant therapy

INTERVENTIONS:
Drug: Pregabalin and venlafaxine concomitant therapy — The control group will only receive an increased dosage of pregabalin and venlafaxine regimen. Each participant will be instructed with the same dose escalation regimen, until they reach the maximal tolerated dose (MTD) or the ceiling dose or the maximum daily recommended dose. The maximum recommended daily dose of pregabalin was 450 mg and venlafaxine was 225 mg.
  Arms: Control group
Drug: Esketamine plus pregabalin and venlafaxine concomitant therapy — The treatment group, in addition to the increased pregabalin and venlafaxine medication dosage regimen, will also receive a single intravenous infusion of esketamine on the day of enrollment. Plasma concentrations of esketamine and its metabolites will be measured at the end of infusion to enable a limited characterization of systemic exposure and to support exploratory exposure-response analyses. Each participant will be instructed with the same dose escalation regimen, until they reach the maximal tolerated dose (MTD) or the ceiling dose or the maximum daily recommended dose. The maximum recommended daily dose of pregabalin was 450 mg and venlafaxine was 225 mg.
  Arms: Treatment group

SUMMARY:
Fibromyalgia is a chronic pain syndrome where current medications have limited efficacy and a slow onset of action. Esketamine shows potential as a rapid-acting analgesic, but previous low-dose studies failed to demonstrate long-term benefits. The efficacy of higher-dose ESK as an adjunctive therapy when standard treatments are insufficient remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients between ages over 18 years with proper cognitive function and language skills for the study;
* Patients diagnosed with FM as defined by the ACR FM diagnostic criteria;
* Patients who have experienced insufficient symptom relief with non-pharmacological treatments and have not previously received recommended pharmacological treatment for FM;
* A score of ≥ 4 on the average pain intensity over 7 days on the numeric rating scale (NRS) at baseline.

Exclusion criteria:

* Patient refusal;
* Inability to sign informed consent;
* Had other secondary FM, this is, hypothyroidism, nutritional deficiency, diabetes mellitus, connective tissue disorder;
* Had psychiatric disorder, this is, schizophrenia and other psychotic disorder, bipolar disorder, or personality disorder;
* Obstructive sleep apnea syndrome or a STOP-Bang score ≥ 3;
* History of treatment with pregabalin and/or venlafaxine for any disease;
* History of treatment with intravenous ketamine or ESK for chronic pain;
* Presence of other painful ailments such as inflammatory rheumatic disease;
* Uncontrolled diabetes, refractory hypertension, malignancies, narrow-angle glaucoma, hyperthyroidism, severe cardiovascular disease or any other contraindications to esketamine;
* History of prescription drug abuse, alcoholism or illicit drug use;
* Pregnant or lactating women;
* Allergic to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
The median pain relief time | At 15 minutes, 1 hour, and 3 hours following termination of treatment, days 1, 3, 5, weeks 1, 2, 4, 8, and 12 for a total of 12 weeks.
  The median pain relief time, defined as the time of 50% decrease in NRS score from baseline. Pain intensity will be measured using the NRS, where 0 indicates no pain, and 10 represents the worst imaginable pain.

SECONDARY OUTCOMES:
Average pain intensity | At the weeks 1, 2, 4, 8, and 12
  The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
Worst pain intensity | at weeks 1, 2, 4, 8, and 12
  The worst pain intensity over the past 24 hours, rated each morning upon awakening and averaged over 7 days. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
Proportion of patients achieving pain reduction at 50% and 30%; | at weeks 1, 2, 4, 8, and 12
  The proportion of patients achieving a ≥ 50% and ≥ 30% reduction in mean baseline pain intensity. The pain intensity will be measured based on NRS, where 0 represents no pain and 10 represents worst pain imaginable.
The maximal tolerated doses of pregabalin and venlafaxine | at weeks 1, 2, 4, 8, and 12
The Revised FM Impact Questionnaire (FIQR) | At the weeks 4, 8, and 12
  The FIQR is used to assessed health status and functional disablity. FIQR is a 21-item self-administered questionnaire, based on symptoms reported within the preceding 7 days. FIQR total score ranges from 0 to 100, with higher values indicating worse health status.
Hospital Anxiety and Depression scale (HADS) | At the weeks 4, 8, and 12
  The HADS is used to assess anxiety (7 items) and depression (7 items). Scores range from 0 to 21 on each subscale, with higher scores indicating worse symptomatology.
The short-form 36 Health Survey (SF-36) | At the weeks 4, 8, and 12
  The SF-36 assesses health-related quality of life, capturing preferences across various health states. It assesses 8 dimensions: physical functioning, physical role limitations due to physical health, bodily pain, general health, vitality, social functioning, emotional role limitations due to emotional problems, and mental health. Scores range from 0 to 100 for each dimension, with higher scores indicating better health status.
Multidimensional Fatigue Inventory (MFI) | At the weeks 4, 8, and 12
  Fatigue is evaluated using the MFI, a 20-item assessment tool with five domains. Higher scores indicate a higher degree of fatigue.
Medical Outcomes Study Sleep Scale (MOS) | At the weeks 4, 8, and 12
  The MOS is a questionnaire comprising 12 items that assess various aspects of sleep using a 6-point ordinal scale (1 indicating permanence and 6 indicating absence).
Plasma concentrations of esketamine and its metabolites at the end of infusion | At the end of esketamine infusion, that is at day 0
Adverse events | Through study completion, an average of 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing 100070, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- See also: Mathieson S, Lin C-WC, Underwood M, Eldabe S. Pregabalin and gabapentin for pain. BMJ. 2020;369:m1315. doi: 10.1136/bmj.m1315 — https://pubmed.ncbi.nlm.nih.gov/32345589/
- See also: Gilron I, Chaparro LE, Tu D, Holden RR, Milev R, Towheed T, et al. Combination of pregabalin with duloxetine for fibromyalgia: a randomized controlled trial. Pain. 2016;157(7):1532-40. doi: 10.1097/j.pain.0000000000000558. — https://pubmed.ncbi.nlm.nih.gov/26982602/
- See also: VanderWeide LA, Smith SM, Trinkley KE. A systematic review of the efficacy of venlafaxine for the treatment of fibromyalgia. J Clin Pharm Ther. 2015;40(1):1-6. doi: 10.1111/jcpt.12216. — https://pubmed.ncbi.nlm.nih.gov/25294655/